CLINICAL TRIAL: NCT06288373
Title: Neoadjuvant Chemoimmunotherapy Combined With Surgery Versus Concurrent Chemoradiotherapy for Locally Advanced Cervical Cancer: a Multicenter Randomized Controlled Clinical Trial
Brief Title: Neoadjuvant Chemoimmunotherapy Versus Concurrent Chemoradiotherapy for LACC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Southwest Hospital, China (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Anhui Provincial Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Qilu Hospital of Shandong University (Other); Beijing Friendship Hospital (Other); Tianjin Medical University General Hospital (Other); West China Second University Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Xiangya Hospital of Central South University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Zhejiang Cancer Hospital (Other); Shengjing Hospital (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Kezhen Li, Prof, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACI-CERV-003; MA-CERVC-II/III-006 (Other Grant/Funding Number: Jiangsu Hengrui Pharmaceuticals Company Ltd.); [2024](S018) (Other: Ethics Committee of Tongji Medical College, HUST)
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer; Locally Advanced Cervical Cancer; Concurrent Chemoradiotherapy; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Cisplatin; Taxes; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab combined neoadjuvant chemotherapy plus radical surgery (Experimental): Patients receive 1 cycle of cisplatin and nab paclitaxel combined neoadjuvant chemotherapy and subsequent 2 cycles of camrelizumab combined neoadjuvant chemotherapy. Based on the tumor size as indicated by MRI, patients who achieve complete response or partial response (CR/PR，RECIST v1.1) will undergo open radical hysterectomy and pelvic lymph node dissection. Patients who show stable disease or progression (SD/PD，v1.1) will proceed directly to concurrent chemoradiotherapy (CCRT).
  Interventions: Drug: Camrelizumab; Drug: Cisplatin; Drug: Nab paclitaxel; Procedure: Radical surgery
- Concurrent Chemoradiotherapy (CCRT) (Active Comparator): Pelvic EBRT + concurrent platinum-containing chemotherapy + brachytherapy
  Interventions: Radiation: external beam radiation therapy (EBRT) + brachytherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q3w (second and third cycles) before radical surgery
  Arms: Camrelizumab combined neoadjuvant chemotherapy plus radical surgery
Drug: Cisplatin — Cisplatin：75-80mg/m2, D1-D2，q3w (3 cycles)，intravenous infusion, administered at a rate of 1mg/min.
  Arms: Camrelizumab combined neoadjuvant chemotherapy plus radical surgery
Drug: Nab paclitaxel — Nab paclitaxel: 260 mg/m2，D1，q3w （3 cycles），intravenous infusion, administered over 30min.
  Arms: Camrelizumab combined neoadjuvant chemotherapy plus radical surgery
Procedure: Radical surgery — Radical surgery
  Arms: Camrelizumab combined neoadjuvant chemotherapy plus radical surgery
Radiation: external beam radiation therapy (EBRT) + brachytherapy — Radiation therapy per standard of care
  Arms: Concurrent Chemoradiotherapy (CCRT)
Drug: Cisplatin — Chemotherapy administered concurrent with radiation therapy，cisplatin 40 mg/m2 IV once per week (QW) for 5 weeks
  Arms: Concurrent Chemoradiotherapy (CCRT)

SUMMARY:
It is a prospective, open-label, randomized, controlled phase II/III clinical trial in which patients with PD-L1-positive FIGO stage IB3, IIA2 and IIB（tumors >4 cm in diameter）will be enrolled and randomly divided into the neoadjuvant chemoimmunotherapy plus surgery group and the CCRT group.

DETAILED DESCRIPTION:
Cervical cancer is the most common gynecological malignancy in China, with locally advanced cervical cancer (LACC) accounting for approximately 37% of cases. Currently, the recommended standard of care for LACC according to international guidelines is concurrent chemoradiotherapy (CCRT). However, the impacts of radiation therapy on patients' quality of life are increasingly being recognized. Additionally, 23.3% to 34.4% of patients still face recurrence or metastasis after treatment, and the 5-year overall survival rate remains around 75%.

Neoadjuvant chemotherapy (NACT) is a chemotherapy regimen used prior to surgery for LACC. NACT followed by radical surgery has a similar overall survival compared to CCRT, but the disease-free survival is relatively lower with NACT. Moreover, 9.8% to 30.6% of patients show poor response to NACT, and over 30% of patients require postoperative adjuvant therapy. These issues significantly limit the application of NACT in LACC.

In recent years, immunotherapy has made significant progress in advanced or recurrent cervical cancer. A phase II clinical trial of combination of PD-1 inhibitors and neoadjuvant chemotherapy showed significant anti-tumor activity and safety. Therefore, based on the preliminary results, this project aims to conduct a multicenter, prospective, randomized controlled clinical trial to further confirm the value of neoadjuvant immunotherapy combined with surgery in LACC. It will be compared with the standard CCRT regimen to explore the differences in clinical efficacy and adverse events between the two groups, providing high-level evidence for the application of neoadjuvant immunotherapy in cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced (2018 FIGO staged IB3, IIA2 and IIB（tumor size> 4cm) ) cervical cancer，staging determined by two physicians of associate seniority or higher after gynecologic examination and imaging evaluation);
2. At least one measurable lesion at baseline according to RECIST 1.1 criteria, with lesion size based primarily on magnetic resonance imaging;
3. Pathologically confirmed diagnosis of cervical cancer, including cervical squamous cell carcinoma, adenocarcinoma (common type), and adenosquamous carcinoma;
4. Positive PD-L1 expression, Combined Positive Score (CPS) ≥1;
5. Patient age ≥18 years and ≤70 years;
6. ECOG score ≤1;
7. Laboratory tests: WBC (white blood cell count) ≥ 3.5×109/L, NEU (neutrophil count) ≥ 1.5×109/L, PLT (platelet count) ≥ 100×109/L, total bilirubin ≤ 1.5 times the upper limit of normal, ALT (alanine aminotransferase) and AST (aspartate aminotransferase) ≤ 1.5 times the upper limit of normal, serum creatinine (BUN) ≤ 1.5 times the upper limit of normal or creatinine clearance ≥ 50 mL/min (calculated using the Cockcroft-Gault formula, the Chronic Kidney Disease Epidemiology Collaboration equation, or the Modification of Diet in Renal Disease equation);
8. Be willing to follow up and good compliance;
9. Be willing to sign the informed consent, including compliance with the requirements and restrictions listed in the informed consent and program；
10. Agree to use effective contraception measures during the trial period and for 5 months after the last dose of pembrolizumab or 6 months after chemotherapy (whichever is longer).

Exclusion Criteria:

1. Any active autoimmune disease or history of autoimmune disease requiring systemic treatment, including but not limited to autoimmune hepatitis, interstitial pneumonitis, uveitis, enterocolitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction, asthma requiring bronchodilator intervention;
2. Prior treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies; known hypersensitivity to any component of the study medication or other monoclonal antibodies;
3. Has a history of human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-DNA ≥ 2000 IU/mL or 104 copies/mL), and hepatitis C (HCV antibody positive, and HCV-RNA above the lower limit of detection of the assay);
4. Receipt of immunosuppressive medications or systemic corticosteroid therapy for immunosuppression (>10 mg/day prednisone or equivalent) within 2 weeks prior to study dosing;
5. Diagnosed with another primary malignancy within 5 years prior to the first use of the investigational drug;
6. Received other investigational drugs/treatments or participated in another clinical trial within 4 weeks prior to randomization. Participation in observational and non-interventional clinical trials is allowed;
7. Pregnant or breastfeeding female patients;
8. Uncontrolled co-morbidities, including but not limited to New York Heart Association (NYHA) class 2 or higher, severe/unstable angina pectoris, myocardial infarction within ≤ 6 months prior to study drug administration, severe arrhythmias requiring medication or intervention; difficult-to-control hypertension; cerebral vascular accidents or brain disorders within ≤ 6 months prior to study drug administration, or individuals with adjudicated abnormal behavioral skills; hematologic disorders: coagulation abnormalities (INR >2. 0, PT>16s), bleeding tendency, or undergoing thrombolytic or anticoagulant therapy; abnormalities in hepatic or renal development or a history of surgery; and development of an active infection requiring systemic anti-infective therapy within 14 days prior to the first dose of study drug;
9. Treatment with a live or attenuated vaccine administered within 4 weeks prior to the first dose of study drug; inactivated seasonal influenza virus vaccine is permitted;
10. Patients with a prior allogeneic bone marrow or solid organ transplant;
11. Drug and/or alcohol abuse;
12. Patients who, in the opinion of the investigator, are unlikely to comply with the procedures, restrictions, and requirements of the study may not be enrolled in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival, PFS | 7 years
  PFS is defined as the time from randomisation to tumor progression, postoperative relaspse or metastasis, or death, which occur first.
Objective Response Rate, ORR | 2 years
  The proportion of patients who had either complete response or partial response, assessed by independent central reviewers according to RECIST, version 1.1.

SECONDARY OUTCOMES:
Overall survival, OS | 7 years
  OS is defined as the time from randomisation to death.
Proportion of patients undergoing radical surgery | 2 years
  Proportion of patients undergoing radical surgery for neoadjuvant chemoimmunotherapy plus surgery group
Pathologic Complete Response | 2 years
  Pathologic complete response (pCR) refers to the absence of invasive/in situ cancer in the cervical and/or lymph nodes.
The surgical complication rate | 2 years
  Intraoperative bleeding, vascular injuries, bladder injuries, rectal injuries, and ureteral injuries were measured by the need for suture repair; occlusive nerve injuries were measured by complete severance, and vascular injuries required documentation of the site of injury. Postoperative complications included: cervical stenosis, cervical insufficiency, ureteral/bladder/rectal/vaginal fistula, internal hemorrhage, pelvic infection, lymphocyst, lymphatic fistula, lower extremity edema, lower extremity venous thrombosis, urinary retention, nerve injury, and bowel obstruction.
Safety and toleraty | 7 years
  The incidence of adverse evetns, severe adverse events; surgery related safety.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Physical Function Score | 7 years
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=not at all to 4=very much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better quality of life. The change from baseline in physical function (EORTC QLQ-C30 Items 1-5) score will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Score | 7 years
  The EORTC QLQ-CX24 is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. The change from baseline in EORTC QLQ-CX24 score will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, Study Chair — Tongji Hospital
Locations (12):
- China (12):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beiing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital (Southwest Hospital), Army Medical University (Third Military Medical University), Chongqing, Chongqing Municipality
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Gansu
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Second People's Hospital of Sichuan (Sichuan Cancer Hospital), Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou Institute of Medicine (HIM), Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No